CLINICAL TRIAL: NCT03766685
Title: A Multicenter, Randomized, Open-Label Study to Evaluate the Safe and Effective Use of the Prefilled Safety Syringe or the Auto-Injector for the Subcutaneous Self-Injection of Bimekizumab Solution by Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Safe and Effective Use of the Prefilled Safety Syringe or the Auto-injector for the Subcutaneous Self-injection of Bimekizumab Solution by Subjects With Moderate to Severe Chronic Plaque Psoriasis (PSO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV0002
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Chronic Plaque Psoriasis
Keywords: Bimekizumab; PSO; Psoriasis; Auto-Injector
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab-SS (Experimental): Subjects will receive assigned bimekizumab dose regimen using a prefilled safety syringe (SS).
  Interventions: Drug: Bimekizumab
- Bimekizumab-AI (Experimental): Subjects will receive assigned bimekizumab dose regimen using an auto-injector (AI).
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: UCB4940; BKZ

SUMMARY:
The purpose of the study is to evaluate the ability of subjects with moderate to severe chronic plaque psoriasis (PSO) to safely and effectively self-inject bimekizumab at study start and 8 weeks after training in self-injection technique using a prefilled safety syringe or an auto-injector.

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfills all inclusion criteria for the PS0014 [NCT03598790] study
* Subject is considered reliable and capable of adhering to the DV0002 protocol (eg, able to understand and complete questionnaires, willing to self-inject, able to use investigational device according to the instructions for use (IFU), and able to adhere to the visit schedule) according to the judgment of the Investigator

Exclusion Criteria:

* Subjects are not permitted to enroll in DV0002 if any of the PS0014 [NCT03598790] study exclusion criteria are met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (39):
- United States (27):
  - Dv0002 946, Phoenix, Arizona
  - Dv0002 910, Bakersfield, California
  - Dv0002 955, San Diego, California
  - Dv0002 943, San Luis Obispo, California
  - Dv0002 967, Santa Monica, California
  - Dv0002 906, Boca Raton, Florida
  - Dv0002 907, Miami, Florida
  - Dv0002 903, Ocala, Florida
  - Dv0002 936, Tampa, Florida
  - Dv0002 941, Alpharetta, Georgia
  - Dv0002 954, Skokie, Illinois
  - Dv0002 900, West Des Moines, Iowa
  - Dv0002 905, Overland Park, Kansas
  - Dv0002 962, Owensboro, Kentucky
  - Dv0002 922, Baton Rouge, Louisiana
  - Dv0002 925, Brighton, Massachusetts
  - Dv0002 917, Troy, Michigan
  - Dv0002 915, St Louis, Missouri
  - Dv0002 901, Portsmouth, New Hampshire
  - Dv0002 908, East Windsor, New Jersey
  - Dv0002 913, New York, New York
  - Dv0002 963, Rochester, New York
  - Dv0002 920, Portland, Oregon
  - Dv0002 929, Portland, Oregon
  - Dv0002 937, Johnston, Rhode Island
  - Dv0002 951, Houston, Texas
  - Dv0002 914, San Antonio, Texas
- Canada (12):
  - Dv0002 672, Edmonton
  - Dv0002 673, Halifax
  - Dv0002 671, Hamilton
  - Dv0002 675, Markham
  - Dv0002 663, Mississauga
  - Dv0002 660, Montreal
  - Dv0002 665, Québec
  - Dv0002 651, Richmond Hill
  - Dv0002 653, Toronto
  - Dv0002 662, Toronto
  - Dv0002 657, Waterloo
  - Dv0002 670, Windsor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sebastian M, Bagel J, Hoepken B, Knapp B, Bicer C, MacPherson M, Langley RG. Single-Injection Options for Administering a 320 mg Dose of Bimekizumab: 2 mL Safety Syringe and Auto-injector. Dermatol Ther (Heidelb). 2025 May;15(5):1113-1134. doi: 10.1007/s13555-025-01366-6. Epub 2025 Mar 29. PMID 40156698
- [Derived] Bagel J, Tatla D, Hellot S, Knapp B, Murphy C, Peterson L, Sebastian M. Bimekizumab Self-Injection Devices: Two Multicenter, Randomized, Open-Label Studies on Self-Administration by Patients With Psoriasis. J Drugs Dermatol. 2022 Feb 1;21(2):162-171. doi: 10.36849/jdd.6274. PMID 35133113
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in December 2018 and concluded in September 2020. This study is a substudy to PS0014 (NCT03598790).
Pre-assignment Details: Participant flow refers to Enrolled Set.
Groups:
- Bimekizumab-SS-1mL 320 mg: Participants self-injected bimekizumab (BKZ) 320 milligrams (mg) solution as a subcutaneous (sc) injection with bimekizumab-Safety Syringe-1 milliliter (mL) (BKZ-SS-1mL) device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on every 4 weeks (Q4W) and every 8 weeks (Q8W) dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml prefilled syringe (PFS) at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16.
- Bimekizumab-AI-1mL 320 mg: Participants self-injected BKZ 320 mg solution as a sc injection with bimekizumab-Auto-Injector-1mL (BKZ-AI-1mL) device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16.
- Bimekizumab-SS-2mL 320 mg: Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-2mL device presentation (ie. 1 self-injection) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 16.
- Bimekizumab-AI-2mL 320 mg: Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-AI-2mL device presentation (ie. 1 self-injection) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 16.
Period: Overall Study
Arm/Group | Bimekizumab-SS-1mL 320 mg | Bimekizumab-AI-1mL 320 mg | Bimekizumab-SS-2mL 320 mg | Bimekizumab-AI-2mL 320 mg
Started | 66 | 68 | 19 | 19
Completed | 65 | 61 | 19 | 18
Not Completed | 1 | 7 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Adverse Event, not fatal | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) consisted of all study participants who received at least 1 dose of bimekizumab by the indicated self-injection investigational device presentation (bimekizumab-SS-1mL SS [SS-s], bimekizumab-AI-1mL SS [SS-a], bimekizumab-SS-2mL SS [SS-s] and bimekizumab-AI-2mL SS [SS-a]). One study participant included in the Enrolled Set did not self-inject at any time during the study and is therefore not included in the Safety Set (SS-s-1mL).
Groups:
- Bimekizumab-SS-1mL 320 mg (SS-s-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the Safety Set (SS) for the 1mL safety syringe (s) device presentation (SS-s-1mL).
- Bimekizumab AI-1mL 320 mg (SS-a-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with bimekizumab-Auto-Injector-1mL (BKZ-AI-1mL) device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the SS for the 1mL auto-injector (a) device presentation (SS-a-1mL).
- Bimekizumab-SS-2mL 320 mg (SS-s-2mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-2mL device presentation (ie. 1 self-injection) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 16. Participants formed the SS for the 2mL safety syringe (s) device presentation (SS-s-2mL).
- Bimekizumab-AI-2mL 320 mg (SS-a-2mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-AI-2mL device presentation (ie. 1 self-injection) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 16. Participants formed the SS for the 2mL auto-injector (a) device presentation (SS-a-2mL).
Arm/Group | Bimekizumab-SS-1mL 320 mg (SS-s-1mL) | Bimekizumab AI-1mL 320 mg (SS-a-1mL) | Bimekizumab-SS-2mL 320 mg (SS-s-2mL) | Bimekizumab-AI-2mL 320 mg (SS-a-2mL) | Total Title
Number analyzed (Participants) | 65 | 68 | 19 | 19 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 0 | 2
  Between 18 and 65 years | 57 | 59 | 16 | 18 | 150
  >=65 years | 7 | 8 | 3 | 1 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (13.4) | 46.8 (14.0) | 50.3 (15.8) | 43.0 (12.4) | 47.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 9 | 9 | 59
  Male | 43 | 49 | 10 | 10 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 2 | 1 | 2 | 7
  Black or African American | 2 | 2 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 2
  White | 60 | 61 | 16 | 16 | 153
  Other or Mixed | 1 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Able to Self-administer Safe and Effective Injections Using the Bimekizumab-safety Syringe (SS)-1mL or the Bimekizumab-auto-injector (AI)-1mL at Week 8, After Training in Self-injection Technique
Description: Safe and effective self-injection was evaluated by the study personnel and was defined as: - Complete dose delivery: Participant self-injected the complete dose of bimekizumab as confirmed by a visual inspection of the bimekizumab-safety syringe (SS) or the bimekizumab-auto-injector (AI) which shows that the investigational medicinal product (IMP) was delivered completely (ie, container is empty), and - No Adverse Device Effects (ADEs) that would preclude continued use of the device for self-injection (ie, no serious ADEs (SADEs) and/or ADEs leading to withdrawal).
Time Frame: Week 8
Population: The Full Analysis Set for device presentation bimekizumab-SS-1mL (FAS-s-1mL) and bimekizumab-AI-1mL (FAS-a-1mL) consisted of all study participants in the SS-s-1mL and SS-a-1mL who self-injected at least 1 dose of bimekizumab using the given device presentation and who had an assessment of self-injection. Here, number of participants were included who were evaluable for the assessment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Bimekizumab-SS-1mL 320 mg (FAS-s-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the Full Analysis Set (FAS) for the 1mL safety syringe (s) device presentation (FAS-s-1mL).
- Bimekizumab -AI-1mL 320 mg (FAS-a-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-AI-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the FAS for the 1mL auto-injector (a) device presentation (FAS-a-1mL).
Arm/Group | Bimekizumab-SS-1mL 320 mg (FAS-s-1mL) | Bimekizumab -AI-1mL 320 mg (FAS-a-1mL)
Number analyzed (Participants) | 63 | 62
percentage of participants | 100 [95.4 to 100] | 100 [95.3 to 100]

2. Primary Outcome: Percentage of Participants Able to Self-administer Safe and Effective Injections Using the Bimekizumab-SS-2mL or the Bimekizumab-AI-2mL at Week 8, After Training in Self-injection Technique
Description: Safe and effective self-injection was evaluated by the study personnel and was defined as: - Complete dose delivery: Participant self-injected the complete dose of bimekizumab as confirmed by a visual inspection of the bimekizumab-SS or the bimekizumab-AI which shows that the IMP is delivered completely (ie, container is empty), and - No ADEs that would preclude continued use of the device for self-injection (ie, no serious ADEs (SADEs) and/or ADEs leading to withdrawal).
Time Frame: Week 8
Population: The Full Analysis Set for device presentation bimekizumab-SS-2mL (FAS-s-2mL) and bimekizumab-AI-2mL (FAS-a-2mL) consisted of all study participants in the SS-s-2mL and SS-a-2mL who self-injected at least 1 dose of bimekizumab using the given device presentation and who had an assessment of self-injection.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Bimekizumab-SS-2mL 320 mg (FAS-s-2mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-2mL device presentation (ie. 1 self-injection) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 16. Participants formed the FAS for the 2mL safety syringe (s) device presentation (FAS-s-2mL).
- Bimekizumab-AI-2mL 320 mg (FAS-a-2mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-AI-2mL device presentation (ie. 1 self-injection) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 2ml PFS at Week 16. Participants formed the FAS for the 2mL auto-injector (a) device presentation (FAS-a-2mL).
Arm/Group | Bimekizumab-SS-2mL 320 mg (FAS-s-2mL) | Bimekizumab-AI-2mL 320 mg (FAS-a-2mL)
Number analyzed (Participants) | 19 | 19
percentage of participants | 100 [85.4 to 100] | 94.7 [77.4 to 99.7]

3. Secondary Outcome: Percentage of Participants Able to Self-administer Safe and Effective Injections Using the Bimekizumab-SS-1mL or the Bimekizumab-AI-1mL at Baseline, After Training in Self-injection Technique
Description: Safe and effective self-injection was evaluated by the study personnel and was defined as: - Complete dose delivery: Participant self-injected the complete dose of bimekizumab as confirmed by a visual inspection of the bimekizumab-SS or the bimekizumab-AI which showed that the IMP was delivered completely (ie, container is empty), and - No ADEs that would preclude continued use of the device for self-injection (ie, no SADEs and/or ADEs leading to withdrawal).
Time Frame: Baseline (the first self-injection visit)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Bimekizumab-SS-1mL 320 mg (FAS-s-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the FAS for the 1mL safety syringe (s) device presentation (FAS-s-1mL).
Arm/Group | Bimekizumab-SS-1mL 320 mg (FAS-s-1mL) | Bimekizumab -AI-1mL 320 mg (FAS-a-1mL)
Number analyzed (Participants) | 64 | 68
percentage of participants | 100 [95.4 to 100] | 97.1 [91.0 to 99.5]

4. Secondary Outcome: Percentage of Participants Able to Self-administer Safe and Effective Injections Using the Bimekizumab-SS-2mL or the Bimekizumab-AI-2mL at Baseline, After Training in Self-injection Technique
Description: Safe and effective self-injection was evaluated by the study personnel and was defined as: - Complete dose delivery: Participant self-injected the complete dose of bimekizumab as confirmed by a visual inspection of the bimekizumab-SS or the bimekizumab-AI which shows that the IMP is delivered completely (ie, container is empty), and - No ADEs that would preclude continued use of the device for self-injection (ie, no SADEs and/or ADEs leading to withdrawal).
Time Frame: Baseline (the first self-injection visit)
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bimekizumab-SS-2mL 320 mg (FAS-s-2mL) | Bimekizumab-AI-2mL 320 mg (FAS-a-2mL)
Number analyzed (Participants) | 19 | 19
percentage of participants | 100 [85.4 to 100] | 100 [85.4 to 100]

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 16
Description: As pre-specified in protocol and SAP, this sub-study collected only specific Adverse Events (AEs) indicated as injection site reactions during selfinjection and investigational device-related AEs - i.e., adverse device effects (ADEs) and serious ADEs, which are reported.Treatment-Emergent (TE)ADEs were defined as AEs related to study device that have a start date on or following the first self-administration of study treatment through the final self-administration of study treatment plus 7 days.
Groups:
- Bimekizumab-SS-1mL 320 mg (SS-s-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-SS-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the SS for the 1mL safety syringe (s) device presentation (SS-s-1mL).
- Bimekizumab AI-1mL 320 mg (SS-a-1mL): Participants self-injected BKZ 320 mg solution as a sc injection with BKZ-AI-1mL device presentation (ie. 2 self-injections) at Baseline and at Week 8 for participants on Q4W and Q8W dosing. For Q4W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 4, 12 and 16. For Q8W dosing, participants were injected by study personnel with 320 mg BKZ using the 1ml PFS at Week 16. Participants formed the SS for the 1mL auto-injector (a) device presentation (SS-a-1mL).
Arm/Group | Bimekizumab-SS-1mL 320 mg (SS-s-1mL) | Bimekizumab AI-1mL 320 mg (SS-a-1mL) | Bimekizumab-SS-2mL 320 mg (SS-s-2mL) | Bimekizumab-AI-2mL 320 mg (SS-a-2mL)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/68 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/68 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/65 | 0/68 | 1/19 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab-SS-1mL 320 mg (SS-s-1mL) (N=65) | Bimekizumab AI-1mL 320 mg (SS-a-1mL) (N=68) | Bimekizumab-SS-2mL 320 mg (SS-s-2mL) (N=19) | Bimekizumab-AI-2mL 320 mg (SS-a-2mL) (N=19)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT03766685/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT03766685/SAP_001.pdf